CLINICAL TRIAL: NCT02342418
Title: Single Dose Pharmacokinetics of Intravenous Tedizolid Phosphate in Morbidly Obese and Age-, Sex-, and Ideal Body Weight-Matched Non-Obese Adults
Brief Title: Single Dose PK of IV Tedizolid Phosphate in Morbidly Obese and Non-Obese Adults
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amit.Pai (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Amit.Pai, Associate Professor, Albany College of Pharmacy and Health Sciences
Organization: Albany College of Pharmacy and Health Sciences (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 14-019
Record Dates: First submitted 2015-01-09; First posted 2015-01-21 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — tedizolid phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Morbidly obese (Active Comparator): The morbidly obese (BMI ≥ 40 kg/m2) arm will be recruited first. Each morbidly obese subject will be matched to a non-obese subject (BMI 18.5-29.9 kg/m2) based on age (± 5 years), sex, and ideal body weight (± 4.6 kg, i.e. ± 5 cm in height). Each group will receive a single dose of tedizolid phosphate 200 mg through a peripheral intravenous catheter.
  Interventions: Drug: Tedizolid phosphate
- Non-obese (Active Comparator): Each non-obese subject will be matched to a morbidly obese subject (BMI 18.5-29.9 kg/m2) based on age (± 5 years), sex, and ideal body weight (± 4.6 kg, i.e. ± 5 cm in height). Each group will receive a single dose of tedizolid phosphate 200 mg through a peripheral intravenous catheter.
  Interventions: Drug: Tedizolid phosphate

INTERVENTIONS:
Drug: Tedizolid phosphate — Each group will receive a single dose of tedizolid phosphate 200 mg through a peripheral intravenous catheter.
  Other Names: Sivextro

SUMMARY:
This is an open label, single-dose, pharmacokinetic study in 9 obese and 9 age-, sex-, ideal body weight- matched non-obese subjects. Qualifying subjects who have completed an informed consent will receive a single intravenous dose of tedizolid with the collection of 11 blood samples over 72 hours post dose.

DETAILED DESCRIPTION:
Subjects will present to the clinical research unit in the morning (approximately 6:30 a.m.) of the dosing day. A urine pregnancy test will be performed to rule out pregnancy prior to administration of the tedizolid phosphate dose to female subjects. The subject's height, total body weight, and vital signs (heart rate, blood pressure, temperature, and respiratory rate) will be recorded. Subjects judged (by study physician) to be healthy enough to participate will proceed with the study procedures.

An 18-20 gauge intravenous peripheral catheter will be inserted into the antecubital vein or a vein in the fore-arm of the non-dominant arm for sequential blood sampling, and an initial predose blood sample (5 mL) will be collected. A minimum of 3-5 mL of blood is required per pharmacokinetic sampling time-point. Each blood collection tube will be pre-labeled with: 1.) study protocol number; 2.) subject study number; 3.) date of collection; 4.) time-point. A 0.9% Sodium Chloride infusion may be run through the peripheral line at 30 to 40 mL per hour to maintain catheter patency for the 12 hour sampling phase. Alternatively, a heparin lock technique will be utilized to maintain intravascular catheter patency.

A single-dose of tedizolid phosphate will be administered as an intravenous infusion (250 mL normal saline) over 1 hour (~8:00 a.m.). The intravenous administration tubing will be flushed with 0.9% Sodium Chloride infusion at 250 mL per hour (to match the tedizolid phosphate rate of infusion) for 10 minutes to ensure complete dose delivery. Blood samples (5 mL) will be collected 0.5 (middle of infusion), 1 (end of infusion), 2, 4, 6, 8, 12, 24, 48, and 72 hours post dose in blood collection tubes. The plasma will be harvested (centrifugation at 4°C) within 60 minutes of collection and stored at -70°C as two aliquots until analysis. The intravascular catheter "dead-space" volume will be discarded prior to blood sample collection by withdrawing 1.5-2 mL from the catheter to ensure no unintentional sample dilution. The intravascular catheter will be removed after the 12 hour sample and the subject will be discharged from the research unit. The subject will return to the research unit for blood sample collection on a daily basis at the following points: 24 (Visit 3), 48 (Visit 4), and 72 hours (Visit 5) after the dose via a peripheral vein needle stick. The exact date and time of blood sample collection will be recorded on case report forms. Each blood sample tube will be inverted and made up-right 5 times to afford mixing of blood with the anticoagulant. Blood samples will be maintained on wet ice and centrifuged at 1200 g for 10 minutes at 4°C within 60 minutes of collection to yield approximately 2 mL of plasma per 5 mL blood collection. The plasma samples will be transferred from the -20°C freezer for storage at -70°C at the end of the sample collection period until analysis.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking or light-smoking (≤ 5 cigarettes per day) volunteers
* Estimated CLcr (Cockcroft-Gault equation) ≥ 90 mL/min
* Female subjects of childbearing potential (CBP) either surgically sterilized, using hormonal contraceptives or an effective barrier method of contraception (diaphragm, cervical cap, condom) or agree to abstain from sex from the time of pre-study screening, during the entire study period and 4 weeks following the study period
* Platelets count ≥ 140,000/mL
* Absolute neutrophil count (ANC) ≥ 1800/mL

Exclusion Criteria:

* History of hypersensitivity reaction to any oxazolidinone
* BMI < 18.5 kg/m2
* Any chronic medical condition requiring pharmacologic therapy
* Transaminases (AST or ALT) > 2.5 x upper limit of normal
* Total bilirubin > 1.5 x upper limit of normal
* Positive urine pregnancy test (if female)
* Abnormal electrocardiogram (ECG) as judged by the study physician
* Unable to tolerate venipuncture and multiple blood draws
* Clinically significant abnormal physical examination defined as a physical finding requiring further clinical work-up
* Unable to independently provide a written informed consent

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-03; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manjunath Pai, PharmD, Principal Investigator — University of Michigan

IPD SHARING:
Plan to Share IPD: No
Summative data have been published

REFERENCES:
- [Result] Pai MP. Pharmacokinetics of Tedizolid in Morbidly Obese and Covariate-Matched Nonobese Adults. Antimicrob Agents Chemother. 2016 Jul 22;60(8):4585-9. doi: 10.1128/AAC.00682-16. Print 2016 Aug. PMID 27185808

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Morbidly Obese | Non-obese
Started | 9 | 10
Completed | 9 | 9
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Morbidly Obese | Non-obese | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Continuous [Median (Full Range); unit: years] | 38 [26 to 50] | 37 [24 to 46] | 37 [24 to 50]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 2 | 2 | 4
Body Mass Index [Median (Full Range); unit: kilogram per square meter] | 43.5 [40.4 to 51.8] | 27.4 [25.4 to 29.1] | 36.1 [25.4 to 51.8]

OUTCOME MEASURES:

1. Primary Outcome: This Outcome Measure is the Tedizolid Area Under the Concentration Time-curve From Time 0 to 72 Hours in Morbidly Obese Subjects and Matched Non-obese Subjects.
Description: The area under the concentration-time curve is measured in units of mg of tedizolid per liter of plasma multiplied by time in hours (hour*mg/L) from time 0 to 72 hours. This comparison was made between the two groups of subjects that included morbidly obese subjects to matched non-obese subjects.
Time Frame: 12 months
Measure: Median (Full Range); unit: hour*milligram/Liter
Arm/Group | Morbidly Obese | Non-obese
Number analyzed (Participants) | 9 | 9
hour*milligram/Liter | 26.0 [18.0 to 42.0] | 27.2 [22.4 to 56.0]
Statistical Analysis 1: Comparison: Morbidly Obese vs Non-obese; Test type: Superiority or Other; p = 0.314, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: This Outcome Measure is the Maximum Plasma Concentration of Tedizolid in Morbidly Obese Subjects Compared to Nonobese Subjects
Description: The maximum concentration or Cmax value is measured in units of milligrams of tedizolid per liter of plasma.This comparison was made between the two groups of subjects that included morbidly obese subjects to matched non-obese subjects.
Time Frame: 12 months
Measure: Mean (Full Range); unit: Milligram per Liter
Arm/Group | Morbidly Obese | Non-obese
Number analyzed (Participants) | 9 | 9
Milligram per Liter | 2.38 [1.28 to 3.99] | 2.96 [2.16 to 5.27]
Statistical Analysis 1: Comparison: Morbidly Obese vs Non-obese; Wilcoxon matched-pair signed-rank test; Test type: Superiority or Other; p = 0.214, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Morbidly Obese | Non-obese
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/10
Other Adverse Events (participants affected / at risk) | 0/9 | 1/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Morbidly Obese (N=9) | Non-obese (N=10)
Intravascular Infiltration (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — During the infusion of the drug into a vein in the drug leaked out to the blood vessel. This is a common side effect that can occur when drugs are administered through a vein.

LIMITATIONS AND CAVEATS:
Most of the participants were below 130 kg and so these data should not be extrapolated to adults above 130 kg.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No